CLINICAL TRIAL: NCT02882698
Title: Performance Analysis in Down Syndrome Through a Maze Game on Mobile Phone
Brief Title: Performance Analysis in Down Syndrome on Mobile Phone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 341/1
Record Dates: First submitted 2016-08-18; First posted 2016-08-30 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Down Syndrome
Keywords: Down syndrome; motor skills; physiotherapy; mobile telephone; exposure to virtual reality therapy
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Down Syndrome Group 1 (Experimental): Acquisition and retention phase on maze A, transfer on maze B and C.
  Interventions: Behavioral: Down Syndrome Group 1
- Down Syndrome Group 2 (Experimental): Acquisition and retention phase on maze C, transfer on maze A and B.
  Interventions: Behavioral: Down Syndrome Group 2
- Typical Development Group 1 (Active Comparator): Control group. Acquisition and retention phase on maze A, transfer on maze B and C.
  Interventions: Behavioral: Typical Development Group 1
- Typical Development Group 2 (Active Comparator): Control group. Acquisition and retention phase on maze C, transfer on maze A and B.
  Interventions: Behavioral: Typical Development Group 2

INTERVENTIONS:
Behavioral: Down Syndrome Group 1 — Acquisition and retention phase on maze A, transfer on maze B and C.
  Arms: Down Syndrome Group 1
Behavioral: Down Syndrome Group 2 — Acquisition and retention phase on maze C, transfer on maze A and B.
  Arms: Down Syndrome Group 2
Behavioral: Typical Development Group 1 — Control group. Acquisition and retention phase on maze A, transfer on maze B and C.
  Arms: Typical Development Group 1
Behavioral: Typical Development Group 2 — Control group. Acquisition and retention phase on maze C, transfer on maze A and B.
  Arms: Typical Development Group 2

SUMMARY:
The game Marble Maze Classic® will be used, in which the participants have to move the mobile phone to conduct a virtual marble through a maze design. The investigators will evaluate 100 individuals (50 with Down Syndrome-DS and 50 with typical development-TD) and divide both with DS and TD into group 1 and 2, where each group consists of 25 participants, with group 2 using a maze design totally opposite to group 1.

DETAILED DESCRIPTION:
The game Marble Maze Classic® will be used, in which the participants have to move the mobile phone to conduct a virtual marble through a maze design. The investigators will evaluate 100 individuals (50 with Down Syndrome-DS and 50 with typical development-TD) and divide both with DS and TD into group 1 and 2, where each group consists of 25 participants, with group 2 using a maze design totally opposite to group 1.

Participants from both SD and TD will be divided into two subgroups: Group 1 (n = 50, consisting of 25 participants in TD and 25 participants in SD) and Group 2 (n = 50, consisting 25 participants in TD and 25 participants in SD), with the design of the maze for group 2 totally opposite to that of group 1 in all stages of the experiment. The use of opposite mazes is necessary to verify that the sequence of movements of the maze path does not influence performance.

To maintain the characteristics of random sampling, where each participant has an equal chance to participate in the groups, The investigators used simple probabilistic random sampling, by conducting the drawing on paper.

PROCEDURES

Individuals will be positioned comfortably in a chair set according to the size necessary, as well as a footrest, so as to stay properly positioned to enable the execution of the task.

Before starting the task, the functioning of the game will be verbally explained, along with a demonstration made by the examiner. The examiner will state that the goal of the game is to get the marble to the end of the maze in the shortest possible time through movements up, down and sideways (supination and pronation of the forearm, flexion and extension of the wrist and fingers). Participants will perform all attempts with the dominant hand (except in intermanual transfer phase) and this task will be repeated several times according to the design of the experiment. In each experiment phase (acquisition, retention and transfer) the execution time will be noted of the entire path from the beginning of the maze until the end point, and in each phase this path has to be performed by a specific amount of repetitions.

To try to match the difficulty of the task, the mazes are customized with paths that require eight basic movements for the virtual marble to reach the target, with two movements of forearm pronation, two supination, two wrist flexion and two extension.

In the design of the learning protocol, the participants have to perform 30 repetitions of the maze task for the acquisition phase with the dominant hand, each group with their own maze. After these 30 repetitions, there was a 5-minute rest period in which the participant is not in contact with the task. Then, 5 repetitions will be performed in the retention phase with the same maze acquisition. For the transfer phase, the participants will perform 15 repetitions divided into 3 blocks of 5 attempts using different maze designs:

* Transfer A: a maze with the path in a different layout to the acquisition (five repetitions);
* Transfer B: the same acquisition maze, however carried out with non-dominant hand (five repetitions);
* Transfer 3: the same acquisition maze with the start-end point of the path reversed (five repetitions).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of DS;
* ability to perform a gripping movement to hold the mobile phone with one of the hands.

Exclusion Criteria:

* presence of comorbidities such as autism or other associated genetic alterations;
* functional disability that impedes the execution of the task or failure of task comprehension after five attempts carried out during the familiarization phase.

Ages: 11 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement of performance | Up to 3 months
  that individuals with DS would be able to adapt to the virtual task using the mobile phone and improve performance with practice in acquisition, as well as maintain the performance in transfer tasks, namely, to change the maze.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Associacao de Pais e Amigos dos Excepcionais de Amparo (APAE), Amparo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided